CLINICAL TRIAL: NCT03413917
Title: Exploration and Determination of Genomic Markers Predictive of Uterine Atony
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 017-356
Record Dates: First submitted 2017-10-31; First posted 2018-01-29 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Uterine Atony
Keywords: genomic markers
MeSH Terms: conditions — Uterine Inertia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — uterine myometrium, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: patients who are admitted for repeat cesarean delivery with bilateral tubal ligation who do not develop uterine atony
  Interventions: Other: Analysis of genomic markers in uterine atony
- Study group: Patients who develop uterine atony either during cesarean delivery or who require surgical management of atony after delivery
  Interventions: Other: Analysis of genomic markers in uterine atony

INTERVENTIONS:
Other: Analysis of genomic markers in uterine atony — No intervention will be performed. We will be analyzing tissue and blood samples only to identify potential association of genomic markers with uterine atony.

SUMMARY:
The primary objective of this study is to determine whether there are markers in the tissue of atonic uteri, and in the patients' plasma that would help identify patients likely to suffer postpartum hemorrhage due to uterine atony. We also will attempt to identify the cause(s) of uterine atony that might suggest mechanisms to prevent and manage it.

DETAILED DESCRIPTION:
Patient will be recruited from those admitted to our Labor and Delivery unit. Ten women will be the control subjects, and these will be selected from patients who are admitted for scheduled cesarean delivery. Ten women will be selected from women who develop uterine atony either following cesarean delivery, or postpartum patients who delivered vaginally but subsequently required surgical management of uterine atony (hysterectomy or uterine saving surgery). From each patient a small amount of uterine muscle will be excised and placed in a fixative, preservative transport medium. Ten cubic centimeters of blood will be drawn from each patient to accompany the tissue. The tissue and blood will be processed and analyzed to identify differences in the tissue and plasma of messenger RNA, micro RNA, long non-coding RNA, and DNA methylation in normal and atonic uterine patients. Statistical analysis of these markers will be performed to determine whether there are significant differences in their expression. It is hoped that differences will be discovered that may be used diagnostically to predict uterine atony, and differences that may suggest the etiology of uterine atony.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* female
* pregnancy over 23 weeks gestation

Exclusion Criteria:

* under 18 years of age
* prisoners
* non-female sex
* cannot provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Our study is to examine genomic markers in uterine atony, thus our subjects must have a uterus.
Study Population: Patients recruited for the study will be pregnant women, 18 years of age or older who are laboring in Labor and Delivery, or who plan to have a scheduled cesarean section.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Identification of genomic markers that can predict uterine atony | 6-12 months
  To extract RNA from serum and uterine tissue samples and use Next Generation miRNA Sequencing followed by quantification of serum miRNA and miRNA isoform expression using TaqMan miRNA assays and NanoString.
Identification of genomic markers that can predict uterine atony (2) | 6-12 months
  Following extraction of miRNA, to use Optical Liquid Stamping technology to analyze various miRNA isoforms in the uterine tissue and serum of subjects with normal uteri compared to atonic uteri.
Identification of genomic markers that can predict uterine atony (3) | 6-12 months
  To isolate DNA using QIAAMp DNA mini kits from uterine tissue and serum samples from subjects with atonic uteri and normal uteri and to then sequence the DNA using HiSeq Genome Analyzer. We will identify the sequence reads using Illumina base-calling software and analyze them using Zymo research proprietary analysis pipeline to identify differences in genomic expression in subjects with normal uteri compared to atonic uteri.

CONTACTS AND LOCATIONS:
Overall Officials: Jack Stecher, MD, Principal Investigator — Baylor Univeristy Medical Center
Locations (1):
- Baylor Univeristy Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toiyama Y, Okugawa Y, Tanaka K, Araki T, Uchida K, Hishida A, Uchino M, Ikeuchi H, Hirota S, Kusunoki M, Boland CR, Goel A. A Panel of Methylated MicroRNA Biomarkers for Identifying High-Risk Patients With Ulcerative Colitis-Associated Colorectal Cancer. Gastroenterology. 2017 Dec;153(6):1634-1646.e8. doi: 10.1053/j.gastro.2017.08.037. Epub 2017 Aug 25. PMID 28847750